CLINICAL TRIAL: NCT06267664
Title: Real-world Effectiveness and Tolerability of Triptans-Ditans-Gepants (TRIDIGEP): an International Prospective Multicentric Cohort Study
Brief Title: Real-world Effectiveness and Tolerability of Triptans-Ditans-Gepants (TRIDIGEP)
Acronym: TRIDIGEP
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, David García Azorín, Principal Investigator, Headache Unit, Department of Neurology, Hospital Clínico Universitario de Valladolid
Other Study IDs: PI-GR-23-3263
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Migraine; Migraine Disorders; Migraine With Aura; Headache Disorders
Keywords: Triptans; Lasmiditan; Gepants
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Headache Disorders | interventions — Tryptamines; lasmiditan; Calcitonin Gene-Related Peptide Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with migraine treated with triptans, Lasmiditan or Gepants: Patients that fulfill the criteria for migraine, according to the International Classification of Headache Disorders, 3rd version treated with triptans, Lasmiditan or Gepants as acute therapies according to their responsible physician criteria under routine clinical practice criteria
  Interventions: Drug: Patients with migraine treated with triptans, Lasmiditan or Gepants

INTERVENTIONS:
Drug: Patients with migraine treated with triptans, Lasmiditan or Gepants — Patients will complete the study information in their smartphones, tablets or computers, using a QR code or a link that will redirect hem to the study questionnaires. RedCap will be used in the study.

SUMMARY:
Migraine is the third most prevalent disease and the leading reason of years lived with disability in the most productive years of the life. Migraine associated disability can be alleviated by acute and preventive treatment. The migraine landscape has changed recently, with the approval of novel acute treatments, including oral Calcitonin gene-related peptide antagonists, the gepants (Rimegepant, Ubrogepant, Zavegepant) and 5-HT-1F antagonists, the Ditans (Lasmiditan). These have joined Triptans as acute "migraine-specific" drugs.

The TRIDIGEP study will be an open-label, multiple attack, prospective cohort study.

This study aims to describe 1) the effectiveness of the acute treatments of migraine attacks in routine clinical practice, 2) the tolerability of the drugs, and 3) to explore potential response and tolerability predictors.

The endpoints recommended by the International Headache Society will be employed, including: 1) Pain freedom; 2) Absence of the most bothersome symptom; 3) Sustained pain freedom; 4) Total freedom from migraine; 5) Headache relief; 6) Duration of attacks; 7) Time lost due to an attack; 8) Need of rescue medication. The study endpoints will be assessed at 2, 8 and 24 hours after the acute drug use. Data will be collected by the patients themselves, with a validated data collection instrument within a RedCap questionnaire, using QR codes.

DETAILED DESCRIPTION:
Introduction Migraine is the third most prevalent disease and the leading reason of years lived with disability in the most productive years of the life. Migraine associated disability can be alleviated by acute and preventive treatment. The migraine landscape has changed in the recent year, with the approval of novel acute treatments, including oral Calcitonin gene-related peptide antagonists, the gepants (Rimegepant, Ubrogepant, Zavegepant) and 5-HT-1F antagonists, the Ditans (Lasmiditan). These have joined Triptans as acute "migraine-specific" drugs.

The reported efficacy of these drugs, assessed by 2-hours pain freedom, is between 25-40% in the case of triptans, 32-39% in the case of Lasmiditan, and 19-35% in the case of gepants. The Achilles tendon of some drugs is tolerability, which may decrease patients' adherence. In the randomized controlled trials (RCTs), the proportion of patients who reported treatment-emergent adverse events (TEAE) was between 2-25% in the case of triptans, 25-40% following Lasmiditan, and 13-17% after Rimegepant. In addition, adverse effects were drug-specific, though (but) luckily only resulted in treatment discontinuation in very few cases. However, due to restrictive eligibility criteria, the population represented in the RCT may differ from the general migraine population.

Aims This study aims to describe 1) the effectiveness of the acute treatments of migraine attacks in routine clinical practice, 2) the tolerability of the drugs, and 3) to explore potential response and tolerability predictors. The endpoints recommended by the International Headache Society will be employed, including: 1) Pain freedom; 2) Absence of the most bothersome symptom; 3) Sustained pain freedom; 4) Total freedom from migraine; 5) Headache relief; 6) Duration of attacks; 7) Time lost due to an attack; 8) Need of rescue medication. The study endpoints will be assessed at 2, 8 and 24 hours after the acute drug use.

This study will facilitate the collection of data from multiple attacks and many patients. The amount of collected data will permit the evaluation of additional outcomes and research questions, by using Big Data and Machine Learning approaches. These questions will include, among others, whether 1) the prompt use of the drug is associated with an increased probability of response; 2) the drug provides a consistent response within several treated attacks in patients; 3) there are any response or no-response predictors; 4) the tolerability of the drug is associated with individual or attack-related factors.

Hypotheses The study hypotheses are that the effectiveness and tolerability of the acute treatments of migraine could differ from the observed efficacy from the randomized clinical trials. The response and tolerability could be related to individual factors or the characteristics of the attack itself.

Study Design The TRIDIGEP study will be an open-label, multiple attack, prospective cohort study. The effectiveness and tolerability of the drugs will be prospectively described by the patients over multiple attacks.

Study Setting The study will be held in multiple headache centers and headache outpatient clinics from the world, including high-income and low-and-middle income countries. All consecutive patients evaluated in the participating sites will be considered for participating in the study. Patients will be informed about the study and invited to participate, if they accept, they will be screened for eligibility. Eligible patients will be trained in the use of the data collection instruments. They will be asked to record the study variables whenever they use the investigated drug products, for at least one attack, but ideally for every attack that they use the drug, ideally for at least five different attacks.

Data will be collected by the patients themselves, with a validated data collection instrument within a RedCap questionnaire. QR codes will be given to the patients to access three different questionnaires: the first one will include the informed consent form signature and the baseline demographic and clinical variables; the second will be for clinical characteristics of the acute migraine attack before the intake of the treatment and the 2-hours effectiveness of the employed drug; and the third one will include the same information in terms of effectiveness and tolerability of the acute drug but 8 and 24 hours after its use. This metodology will reflect how the different drugs are really used, so that factors that might be associated with a better or worse response will also be analyzed. Thus, the study will produce real-world data from many of them, and the benefits of the study will multiply, since data from several drugs will be collected in a standardized way, allowing comparative analyses.

Eligibility criteria Patients will be included if they 1) fulfill the criteria for migraine, according to the International Classification of Headache Disorders, 3rd version; 2) are treated with triptans, Lasmiditan or Gepants as acute therapies according to their responsible physician criteria under routine clinical practice criteria; 3) have a smartphone, tablet, or computer with an internet connection; 4) accept to participate and sign the informed consent form. Patients will be excluded if they 1) have a concomitant use of opioids, barbiturates, or ergot derivates; 2) have major cognitive or psychiatric disorders; 3) are unable to describe the result of the employed drug or have an insufficient proficiency of the local languages.

Variables The study will include demographic variables, prior medical history and clinical variables related with the treated migraine attacks. Demographic variables will include sex, date of birth, height, and weight. Clinical baseline variables will include the type of migraine, the number of headache and migraine days per month, on average, in the preceding three months, the presence of aura, the prior or current use of preventive medications, and the presence of comorbidities. The studied comorbidities will include arterial hypertension, diabetes, hyperlipidemia, smoking or former smoking habit, alcohol misuse; any disorder, including cardiovascular, pulmonary, neurological, neurosurgical, gastrointestinal, hepatic, kidney, otologic, endocrinologic, dermatologic, hematologic, allergy, immunological, oncological or psychiatric systems, including depression, anxiety, insomnia or others.

The information that will be collected related to the headache episode will include the presence of aura prior to the attack, the time when the headache started, and the moment when the drug was used, localization and quality of the pain, headache intensity, and the presence of associated symptoms, including photophobia, phonophobia, osmophobia, worsening by routine physical activity, nausea, vomiting, cranial autonomic symptoms, blurred vision or other symptoms. Patients will select the most bothersome symptom. The employed drug, including the dose and timing, will be assessed.

The clinical variables regarding effectiveness and tolerability will be assessed 2, 8 and 24 hours after drug intake. Effectiveness variables will include the headache intensity, and the presence of associated symptoms, using the same list, at the baseline and over the three time-points. The ability of functioning at the same time-points will be evaluated. Tolerability will be asked by an open question with a free-text response first, and afterwards, a list of possible AEs will be provided, including cutaneous rash, tiredness, gastrointestinal disturbances, constipation, somnolence, nausea, dizziness, vertigo, unsteadiness, sexual dysfunction, chest discomfort, weakness, reduced physical capacity, paresthesia, tingling, palpitations, bradycardia, tachycardia, blurred vision, and others. If patients report any of the listed Aes, a question regarding whether the symptom began after the drug intake or if it was present prior to the drug use will appear. The total duration of the headache, the time lost due to an attack, and the Global Impression of Change will be evaluated at 24 hours.

Data sources / measurements Patients will complete the study information in their smartphones, tablets or computers, using a QR code or a link that will redirect hem to the study questionnaires. RedCap will be used in the study. The questionnaires will be translated into the local languages.

Bias The Newcastle-Ottawa scale and the Risk of Bias in Non-randomized Studies of Interventions (ROBINS-I) criteria have been revised in the study design phase. Regarding patient selection, case definition will be based on the ICHD-3 criteria, cases will be representative of the entire migraine population, and they will act as their own controls, since the study will compare the situation before-after the drug intake.

The outcomes will be assessed with a record linkage through RedCap, and an independent statistician will assess them, blind to the participant's records. The follow-up will be long enough for the outcomes to occur, for 24-hours.

The study cohort will be followed-up adequately, with a complete follow-up. In case that patients are lost to follow-up, their characteristics will be described, and the reasons for patients lost will be provided.

None of the baseline variables will predict the intervention received.

Study size There is no sample size estimation, as we aim to enroll as many patients as possible. The aim is to surpass the sample sizes from the RCTS, which ranged between 200-1500 patients

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria for migraine, according to the International Classification of Headache Disorders, 3rd version;
* Treatment with triptans, Lasmiditan or Gepants as acute therapies according to their responsible physician criteria under routine clinical practice criteria;
* Participant have a smartphone, tablet, or computer with an internet connection;
* Participant accept to participate and sign the informed consent form

Exclusion Criteria:

* Patient have a concomitant use of opioids, barbiturates, or ergot derivates;
* Participant have major cognitive or psychiatric disorder;
* Participants are unable to describe the result of the employed drug
* Participants have an insufficient proficiency of the local languages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients with migraine, according to the International Headache Society criteria. Eligible patients will be trained in the use of the data collection instruments. They will be asked to record the study variables whenever they use the investigated drug products, for at least one attack, but ideally for every attack that they use the drug, ideally for at least five different attacks.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain freedom at 2 hours | Two hours after treatment intake
  The percentage of subjects who become pain free at two hours after treatment, before the use of any rescue medication
Absence of the most bothersome symptom | Two hours after treatment intake
  Absence of the most bothersome migraine-asso- ciated symptom at 2 hours after treatment

SECONDARY OUTCOMES:
Pain freedom at 8 hours | Eight hours after treatment intake
  The percentage of subjects who become pain free at eight hours after treatment, before the use of any rescue medication
Pain freedom at 24 hours | 24 hours after treatment intake
  The percentage of subjects who become pain free at 24 hours after treatment, before the use of any rescue medication
Sustained pain freedom | Twenty-four hours after treatment intake
  percentage of subjects who are pain free at 2 hours with no use of rescue medication or relapse within 24 hours of the initial treatment.
Total freedom from migraine at 2 hours | Two hours after treatment intake
  Percentage of subjects who report Freedom from headache and any migraine- associated symptoms at two hours
Total freedom from migraine at 8 hours | Eight hours after treatment intake
  Percentage of subjects who report Freedom from headache and any migraine- associated symptoms at eight hours
Total freedom from migraine at 24 hours | Twenty-four hours after treatment intake
  Percentage of subjects who report Freedom from headache and any migraine- associated symptoms at 24 hours
Headache relief at 2 hours | Two hours after treatment intake
  Percentage of subjects who report decrease in headache pain from moderate or severe at baseline to mild or none at 2 hours after treatment and before taking any rescue medication
Headache relief at 8 hours | Eight hours after treatment intake
  Percentage of subjects who report decrease in headache pain from moderate or severe at baseline to mild or none at 2 hours after treatment and before taking any rescue medication
Headache relief at 24 hours | 24 hours after treatment intake
  Percentage of subjects who report decrease in headache pain from moderate or severe at baseline to mild or none at 2 hours after treatment and before taking any rescue medication
Time to meaningful relief | 24 hours after treatment intake
  Number of minutes between the acute drug intake and the presence of meaningful relief
Time to pain freedom | 24 hours after treatment intake
  Number of minutes between the acute drug intake and the presence of pain freedom
Time to migraine freedom | 24 hours after treatment intake
  Number of minutes between the acute drug intake and the presence of migraine freedom
Need of rescue medication at 2 hours | 2 hours after treatment intake
  The percentage of patients taking rescue medication 2 hours after intake of the drug
Need of rescue medication at 8 hours | 8 hours after treatment intake
  The percentage of patients taking rescue medication 8 hours after intake of the drug
Need of rescue medication at 24 hours | 24 hours after treatment intake
  The percentage of patients taking rescue medication 24 hours after intake of the drug
Tolerability of the drugs | 24 hours after the treatment intake
  To describe the frequency and type of adverse events
Response predictors at 2 hours | Assessed at 2 hours after the acute drug use.
  To evaluate which demographic and clinical variables are associated with a higher probability of response at 2 hours
Response predictors at 24 hours | Assessed at 24 hours after the acute drug use.
  To evaluate which demographic and clinical variables are associated with a higher probability of response at 24 hours
Tolerability predictors | Assessed at 24 hours after the acute drug use.
  To explore which demographic and clinical variables are associated with the presence of any adverse effect
Time lost due to an attack | 24 hours after the acute drug use
  Number of minutes that the patients was not able to work / act normally due to the headache and associated symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be shared upon reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] VanderPluym JH, Halker Singh RB, Urtecho M, Morrow AS, Nayfeh T, Torres Roldan VD, Farah MH, Hasan B, Saadi S, Shah S, Abd-Rabu R, Daraz L, Prokop LJ, Murad MH, Wang Z. Acute Treatments for Episodic Migraine in Adults: A Systematic Review and Meta-analysis. JAMA. 2021 Jun 15;325(23):2357-2369. doi: 10.1001/jama.2021.7939. PMID 34128998
- [Background] Agostoni EC, Barbanti P, Calabresi P, Colombo B, Cortelli P, Frediani F, Geppetti P, Grazzi L, Leone M, Martelletti P, Pini LA, Prudenzano MP, Sarchielli P, Tedeschi G, Russo A; Italian chronic migraine group. Current and emerging evidence-based treatment options in chronic migraine: a narrative review. J Headache Pain. 2019 Aug 30;20(1):92. doi: 10.1186/s10194-019-1038-4. PMID 31470791
- [Background] Macone AE, Perloff MD. Triptans and migraine: advances in use, administration, formulation, and development. Expert Opin Pharmacother. 2017 Mar;18(4):387-397. doi: 10.1080/14656566.2017.1288721. Epub 2017 Feb 14. PMID 28129702
- [Background] Phebus LA, Johnson KW, Zgombick JM, Gilbert PJ, Van Belle K, Mancuso V, Nelson DL, Calligaro DO, Kiefer AD Jr, Branchek TA, Flaugh ME. Characterization of LY344864 as a pharmacological tool to study 5-HT1F receptors: binding affinities, brain penetration and activity in the neurogenic dural inflammation model of migraine. Life Sci. 1997;61(21):2117-26. doi: 10.1016/s0024-3205(97)00885-0. PMID 9395253
- [Background] Goadsby PJ, Edvinsson L, Ekman R. Release of vasoactive peptides in the extracerebral circulation of humans and the cat during activation of the trigeminovascular system. Ann Neurol. 1988 Feb;23(2):193-6. doi: 10.1002/ana.410230214. PMID 2454066
- [Background] Doods H, Hallermayer G, Wu D, Entzeroth M, Rudolf K, Engel W, Eberlein W. Pharmacological profile of BIBN4096BS, the first selective small molecule CGRP antagonist. Br J Pharmacol. 2000 Feb;129(3):420-3. doi: 10.1038/sj.bjp.0703110. PMID 10711339
- [Background] Yao G, Yu T, Han X, Mao X, Li B. Therapeutic effects and safety of olcegepant and telcagepant for migraine: A meta-analysis. Neural Regen Res. 2013 Apr 5;8(10):938-47. doi: 10.3969/j.issn.1673-5374.2013.10.009. PMID 25206386
- [Background] Luo G, Chen L, Conway CM, Denton R, Keavy D, Signor L, Kostich W, Lentz KA, Santone KS, Schartman R, Browning M, Tong G, Houston JG, Dubowchik GM, Macor JE. Discovery of (5S,6S,9R)-5-amino-6-(2,3-difluorophenyl)-6,7,8,9-tetrahydro-5H-cyclohepta[b]pyridin-9-yl 4-(2-oxo-2,3-dihydro-1H-imidazo[4,5-b]pyridin-1-yl)piperidine-1-carboxylate (BMS-927711): an oral calcitonin gene-related peptide (CGRP) antagonist in clinical trials for treating migraine. J Med Chem. 2012 Dec 13;55(23):10644-51. doi: 10.1021/jm3013147. Epub 2012 Nov 15. PMID 23153230
- [Background] Moreno-Ajona D, Villar-Martinez MD, Goadsby PJ. New Generation Gepants: Migraine Acute and Preventive Medications. J Clin Med. 2022 Mar 16;11(6):1656. doi: 10.3390/jcm11061656. PMID 35329982
- [Background] Diener HC, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Mandrekar J; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition. Cephalalgia. 2019 May;39(6):687-710. doi: 10.1177/0333102419828967. Epub 2019 Feb 26. PMID 30806518
- [Background] Ferrari MD, Roon KI, Lipton RB, Goadsby PJ. Oral triptans (serotonin 5-HT(1B/1D) agonists) in acute migraine treatment: a meta-analysis of 53 trials. Lancet. 2001 Nov 17;358(9294):1668-75. doi: 10.1016/S0140-6736(01)06711-3. PMID 11728541
- [Background] Kuca B, Silberstein SD, Wietecha L, Berg PH, Dozier G, Lipton RB; COL MIG-301 Study Group. Lasmiditan is an effective acute treatment for migraine: A phase 3 randomized study. Neurology. 2018 Dec 11;91(24):e2222-e2232. doi: 10.1212/WNL.0000000000006641. Epub 2018 Nov 16. PMID 30446595
- [Background] Goadsby PJ, Wietecha LA, Dennehy EB, Kuca B, Case MG, Aurora SK, Gaul C. Phase 3 randomized, placebo-controlled, double-blind study of lasmiditan for acute treatment of migraine. Brain. 2019 Jul 1;142(7):1894-1904. doi: 10.1093/brain/awz134. PMID 31132795
- [Background] Lipton RB, Croop R, Stock EG, Stock DA, Morris BA, Frost M, Dubowchik GM, Conway CM, Coric V, Goadsby PJ. Rimegepant, an Oral Calcitonin Gene-Related Peptide Receptor Antagonist, for Migraine. N Engl J Med. 2019 Jul 11;381(2):142-149. doi: 10.1056/NEJMoa1811090. PMID 31291516
- [Background] Croop R, Goadsby PJ, Stock DA, Conway CM, Forshaw M, Stock EG, Coric V, Lipton RB. Efficacy, safety, and tolerability of rimegepant orally disintegrating tablet for the acute treatment of migraine: a randomised, phase 3, double-blind, placebo-controlled trial. Lancet. 2019 Aug 31;394(10200):737-745. doi: 10.1016/S0140-6736(19)31606-X. Epub 2019 Jul 13. PMID 31311674
- [Background] Martinez-Pias E, Garcia-Azorin D, Minguez-Olaondo A, Trigo J, Sierra A, Ruiz M, Guerrero AL. Triptanophobia in migraine: A case-control study on the causes and consequences of the nonuse of triptans in chronic migraine patients. Expert Rev Neurother. 2021 Jan;21(1):123-130. doi: 10.1080/14737175.2021.1842733. Epub 2020 Nov 2. PMID 33111580
- [Background] Thorlund K, Toor K, Wu P, Chan K, Druyts E, Ramos E, Bhambri R, Donnet A, Stark R, Goadsby PJ. Comparative tolerability of treatments for acute migraine: A network meta-analysis. Cephalalgia. 2017 Sep;37(10):965-978. doi: 10.1177/0333102416660552. Epub 2016 Aug 12. PMID 27521843
- [Background] Ashina M, Reuter U, Smith T, Krikke-Workel J, Klise SR, Bragg S, Doty EG, Dowsett SA, Lin Q, Krege JH. Randomized, controlled trial of lasmiditan over four migraine attacks: Findings from the CENTURION study. Cephalalgia. 2021 Mar;41(3):294-304. doi: 10.1177/0333102421989232. Epub 2021 Feb 4. PMID 33541117
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Result] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- See also: European Medicines Agency: Vydura: EPAR - Medicine Overview. Publicado el 11.05.2022 — https://www.ema.europa.eu/documents/overview/vydura-epar-medicine-overview_en.pdf
- See also: European Medicines Agency: Rayvow: EPAR - Medicine Overview. Publicado el 03.10.2022 — https://www.ema.europa.eu/documents/overview/rayvow-epar-medicine-overview_en.pdf
- See also: Santos Lasaosa S, Pozo Rosich P. Manual de Práctica Clínica en Cefaleas. Recomendaciones Diagnóstico- Terapéuticas de la Sociedad Española de Neurología 2020. Ediciones SEN. ISBN: 978-84-18420-19-1. — https://www.sen.es/pdf/2020/ManualCefaleas2020.pdf